CLINICAL TRIAL: NCT06703723
Title: Effect of Cryopreservation on SARS-CoV-2 Semen Samples: Influence of Two Different Cryopreservation Procedures Evaluated After Thawing
Brief Title: Impact of Cryopreservation Methods on Post-Thaw SARS-CoV-2 in Semen Samples
Acronym: SEM-COV-19
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 230879
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: COVID 19
Keywords: sars-cov-2; semen cryopreservation; male reproductive health; viral contamination; inflammation
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Semen samples of individuals that have been exposed to SARS-CoV-2 infection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Male subjects, aged 18-50 requiring a semen fluid evaluation. • Positive IgG serological test result
- Healthy: Healthy

SUMMARY:
Cryopreservation of seminal fluid or spermatozoa from epididymary and testicular retrieval represents a crucial tool in managing conditions of permanent or temporary infertility, as well as in cases of secretory and excretory azoospermia. These pathologies often affect young men and children, making it essential to maintain fertility through cryopreservation methods such as vitrification or two-step cryopreservation of human semen.

The burden of the SARS-CoV-2 virus has rapidly evolved. SARS-CoV-2 causes respiratory, cardiovascular, digestive, and urinary infections, yet no studies have explored its effects on the reproductive system. Recent findings confirm the expression of the virus receptor (ACE2) on certain testicular cells, including Sertoli cells, Leydig cells, and spermatogonia, which could significantly impact fertility and cryopreservation practices.

This study aims to utilize semen samples from individuals exposed to SARS-CoV-2 infection to perform two different cryopreservation procedures, evaluating virus behavior and effects. The objective is to determine whether it is safer to cryopreserve the entire volume of the sample or perform gradient separation to isolate the virus from spermatozoa, potentially establishing a new cryopreservation protocol specific to SARS-CoV-2.

DETAILED DESCRIPTION:
The pandemic caused by SARS-CoV-2 ranks among the most devastating events in recent history. Limited knowledge exists regarding the characteristics and behavior of this beta coronavirus, particularly its potential impact on reproductive medicine. Questions remain about the presence of the virus in seminal fluid and whether male semen could serve as a transmission route. Additionally, concerns exist about the virus impairing male reproductive potential through fever or the "cytokine storm" triggered by the immune response.

No current evidence confirms whether SARS-CoV-2 can survive semen cryopreservation, though other viruses, such as influenza, have demonstrated survival in liquid nitrogen freezing. Semen cryopreservation is a critical fertility preservation strategy for conditions like cancers, autoimmune diseases, or cryptorchidism. The contamination of cryopreserved semen by SARS-CoV-2 could turn such samples into hazardous viral reservoirs.

The study aims to investigate the presence of the virus in semen, identify cells expressing viral receptors ACE2 and TMPRSS2, and evaluate the virus's direct and indirect effects on male reproductive capacity. Objectives include determining if SARS-CoV-2 survives cryopreservation procedures and identifying optimal methods to ensure virus-free cryopreserved semen while separating infected material from male gametes.

The study will recruit 20 men exposed to SARS-CoV-2 and 20 control subjects, all treated at the Humanitas Fertility Center, Department of Gynecology, at the Humanitas Research Hospital. Each participant will provide a semen sample for evaluation. This observational study will not involve clinical interventions or alter regular diagnostic procedures.

Participants undergoing routine tests for medically assisted reproduction and deemed eligible after completing an anamnesis questionnaire will be included. Samples will be processed in the Mucosal Immunology and Microbiota Unit at the Humanitas Clinical Institute.

Using cell biology, molecular biology, and flow cytometry techniques, the study will assess viral contamination, receptor expression in spermatozoa, and inflammatory cytokine levels in seminal fluid after two cryopreservation methods: slow two-step freezing and vitrification. Analyses will cover unprocessed semen and samples exposed in vitro to SARS-CoV-2 under BSL3 conditions.

Additionally, the cellular fraction of semen, including granulocytes, lymphocytes, round cells, and spermatozoa, will undergo phenotype and activation state characterization. The study will evaluate viral contamination in cryopreserved semen and assess the effectiveness of protocols designed to separate infected material from male gametes.

ELIGIBILITY:
Inclusion Criteria:

Patient population inclusion criteria:

* • Male subjects, aged 18-50 requiring a semen fluid evaluation.

  * Positive IgG serological test result performed not more than 3 months before recruitment
  * Signed informed consent
  * Anamnestic test compilation

Control subject inclusion criteria:

* Male subjects, aged 18-50 requiring a semen fluid evaluation.
* Negative IgG serological test result performed within the last month
* Signed informed consent
* Anamnestic test compilation

Exclusion Criteria:

* Patient population exclusion criteria:

  * Severe male Factor (azoospermia and <200,00 sperm per ejaculate)
  * Fever (>38.5 C) in the 60 days before enrollment
  * Treated with antibiotic at the time of enrolment or two months before enrolment
  * Treated with cortisone at the time of enrolment or two months before enrolment

Control subject population exclusion criteria:

* Severe male Factor (azoospermia and <200,00 sperm per ejaculate)
* Fever (>38.5 C) in the 60 days before enrolment
* Known history of SARS-CoV-2 infection
* Treated with antibiotic at the time of enrolment or two months before enrolment
* Treated with cortisone at the time of enrolment or two months before enrolment

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male, since we collect semen samples
Study Population: To analyze the effect of the two cryopreservation methods (slow freezing in two stages and vitrification) on semen samples, we propose to include 20 patients who have been exposed to SARS-CoV-2 infection and 20 control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
nvestigation of ACE2 and TMPRSS2 mRNA Expression on Spermatozoa in SARS-CoV-2 Infected Semen Samples | through study completion, an average of 1 year
  investigate the presence of the mRNA encoding ACE2 and TMPRSS2 on spermatozoa of SARS-CoV-2 semen samples

SECONDARY OUTCOMES:
Impact of Cryopreservation Methods on the Presence of Viral RNA in SARS-CoV-2 Infected Semen: A Comparison of Two-Step Cryogenic Freezing and Vitrification | through study completion, an average of 1 year
  The primary outcome of the study will be to investigate the presence of viral RNA in semen samples after cryopreservation using two-step cryogenic freezing and vitrification methods.
valuation of the Presence of the SARS-CoV-2 Viral Genome in Semen Samples" | through study completion, an average of 1 year
  evaluating the presence of the viral genome
Immune profiling | through study completion, an average of 1 year
  Immune activation compared to controls

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided